CLINICAL TRIAL: NCT04232748
Title: Clinical Significance of Change in Body Weight During Treatment of Advanced Colorectal Cancer Patients - A Pilot Study
Brief Title: Change in Body Weight During Treatment of Advanced Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Shing Fung Lee, Resident Specialist, Tuen Mun Hospital
Other Study IDs: NTWC/CREC/18027
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cancer, Colorectal; Chemotherapy Effect; Weight Loss; Prognosis
Keywords: cancer; survival; chemotherapy; weight
MeSH Terms: conditions — Colorectal Neoplasms; Weight Loss; Neoplasms; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stage IV colorectal cancer: stage IV colorectal cancer on first line systemic treatment are observed for the trend of weight change and treatment outcomes
  Interventions: Drug: first line systemic treatment for colorectal cancer

INTERVENTIONS:
Drug: first line systemic treatment for colorectal cancer — systemic chemotherapy (capecitabine or fluorouracil, oxaliplatin or irinotecan, with or without biological agents including cetuximab, bevacizumab, or panitumumab.

SUMMARY:
Colorectal cancer (CRC) is a significant and growing health burden in Hong Kong. According to data from Hong Kong Cancer Registry, CRC ranked the first in incidence and the second in mortality, with around 5,000 new cases diagnosed and more than 2,000 cancer-related mortality in 2014. The investigators aim to evaluate the association between serial weight change during first line treatment and outcomes in patients with metastatic CRC.

DETAILED DESCRIPTION:
Studies have suggested that exposure to a greater number of chemotherapeutic agents is associated with better survival in metastatic colorectal cancer.

Multiple factors might affect body weight during treatment. Cancer-related symptoms can impair quality of life and appetite. Cachexia syndrome affects around 50% of colon cancer patients and is characterized by cancer-induced catabolism with involuntary weight loss (fat and muscle), patients have increased lipolysis and change in skeletal muscle metabolism, including increased energy expenditure at rest and protein degradation, and decreased protein synthesis. Besides these disease factors, treatment related side effects are common causes of weight loss, such as inability to ingest or digest food effectively due to nausea, vomiting, and malaise. Based on these factors and the hypotheses between tumour control and weight gain, monitoring the serial weight change can have practical value.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of colorectal origin
* Stage IV disease with systemic treatment
* Estimated life expectancy >3 months
* Adequate organ functions

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status 3 or above
* Pregnancy
* Human immunodeficiency virus infection and acquired immune deficiency syndrome (HIV/AIDS)
* Past medical history of another cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single institutional cohort of stage IV (advanced) colorectal cancer patients who undergo systemic treatments.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of start of anti-cancer treatment until the date of first documented progression (assessed by physical examination, imaging, or blood biomarkers) or date of death from any cause, whichever came first, assessed up to 60 months
  Survival time from start of anti-cancer treatment until disease progression, or death from disease, or loss of follow-up
Overall survival | From date of start of anti-cancer treatment until the date of death from any cause (assessed by physical examination, imaging, or blood biomarkers), assessed up to 60 months
  Survival time from start of anti-cancer treatment until death from any cause, or loss of follow-up

SECONDARY OUTCOMES:
Chemotherapy dose change | from start of first-line anti-cancer treatment until completion, assessed by clinical assessment up to 60 months
  Chemotherapy dose change (in percentage change)
Chemotherapy interruption | from start of first-line anti-cancer treatment until completion, assessed by clinical assessment up to 60 months
  Chemotherapy dose interruption (in percentage change)

CONTACTS AND LOCATIONS:
Overall Officials: Shing Fung Lee, MBBS, M Sc, Principal Investigator — Department of Clinical Oncology, Tuen Mun Hospital, Hong Kong
Locations (1):
- Department of Clinical Oncology, Tuen Mun Hospital, Tuen Mun, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Study Protocol (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04232748/Prot_000.pdf